CLINICAL TRIAL: NCT01790581
Title: Balance Training vs. Balance Training w/ STARS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Charlotte (Other)
Collaborators: Mid-Atlantic Athletic Trainers' Association (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: UNCC12-09-16
Record Dates: First submitted 2013-02-08; First posted 2013-02-13 (Estimated); Results first posted 2014-12-24 (Estimated); Last update posted 2017-07-11 (Actual); Status verified 2017-07

CONDITIONS: Ankle (Ligaments); Instability (Old Injury)
Keywords: Chronic Ankle Instability

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Balance Training (Active Comparator)
  Interventions: Behavioral: Balance Training
- Balance Training w/ STARS (Experimental)
  Interventions: Behavioral: Balance Training; Behavioral: STARS

INTERVENTIONS:
Behavioral: Balance Training — This is a 4-week supervised balance training program that has been previously validated in those with CAI by improving subjective and objective measures of function. During the 4-week program, subjects will complete three 20-25 minute sessions a week for a total of twelve supervised training sessions. The specific exercises and repetitions that will be performed per training session will include: 1) hop to stabilization (10 repetitions per direction), 2) hop to stabilization and reach (5 repetitions per direction), 3) unanticipated hop to stabilization (3 repetitions), 4) progressive single limb stance balance activities (3 repetitions), and 5) progressive single limb stance activities with eyes closed (3 repetitions).
Behavioral: STARS — The STARS intervention will consist of 4 unique sensory-targeted interventions: calf stretching, ankle joint traction, anterior/posterior ankle joint mobilizations, and plantar massage. These four techniques target 3 types of sensory pathways (musculotendinous, articular, and plantar cutaneous, respectively) and will be applied in the same order for all treatment sessions: 1) 60-second calf stretch, 2) 30-second ankle traction, 3) 30-second mobilization, 4) 2-minute plantar massage, 5) 30-second ankle traction, and 6) 30-second mobilization.
  Arms: Balance Training w/ STARS

SUMMARY:
Chronic Ankle Instability (CAI) is a health condition that results in repeated ankle sprains and other residual impairments. CAI has been linked to many different causative factors including sensory and motor deficits that affect the global function of the sensorimotor system as well as the patient. Over the past 20 years, strong evidence has been generated to support balance training as an effective intervention strategy in the CAI population. Unfortunately, most investigations have focused solely on maximizing motor output through balance training, while ignoring the full spectrum of sensorimotor dysfunction associated with CAI. There may be advantageous sensory-targeted interventions that augment the effects of balance training and lead to greater enhancements of functional outcomes for CAI. However, this possibility has not been systematically explored. Sensory-targeted ankle rehabilitation strategies (STARS), such as joint mobilization and plantar massage have resulted in improved sensorimotor function in those with CAI. However, only a single STARS (i.e. stochastic resonance) has been investigated in combination with balance training. While the combined effects were greater than those of balance training alone, stochastic resonance requires relatively expensive equipment that is not commercially available. Thus, the purpose of this investigation is to test the hypothesis that combining low cost STARS (e.g. plantar massage and joint mobilizations) with balance training will result in greater sensorimotor and functional improvements in those with CAI than balance training alone.

ELIGIBILITY:
Inclusion Criteria:

* Males and females between the ages of 18 and 35.
* A history of at least one episode of "giving way" within the past 3 months.
* Answering 4 or more questions of "Yes" on the Ankle Instability Instrument (AII).
* Score of <90% on the self-reported Foot and Ankle Ability Measure (FAAM).
* Score of <80% on the FAAM Sport.

Exclusion Criteria:

* Failing to meet the inclusion criteria.
* Known balance and vision problems.
* Acute lower extremities and head injuries that occurred <6 weeks ago.
* Chronic musculoskeletal conditions known to affect balance.
* A history of ankle surgeries to fix internal derangements.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2013-01; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Erik A Wikstrom, PhD, Principal Investigator — University of North Carolina at Charlotte
Locations (1):
- University of North Carolina at Charlotte, Charlotte, North Carolina, United States

REFERENCES:
- [Background] McKeon PO, Ingersoll CD, Kerrigan DC, Saliba E, Bennett BC, Hertel J. Balance training improves function and postural control in those with chronic ankle instability. Med Sci Sports Exerc. 2008 Oct;40(10):1810-9. doi: 10.1249/MSS.0b013e31817e0f92. PMID 18799992
- See also: Link to the laboratory in which the research is being conducted — http://kinesiology.uncc.edu/research-and-scholarship/biodynamics-research-laboratory

RESULTS

PARTICIPANT FLOW:
Groups:
- Balance Training w/ STARS: Balance Training: This is a 4-week supervised balance training program. During the 4-week program, subjects will complete three 20-25 minute sessions a week for a total of twelve supervised sessions. Exercises and repetitions per training session will include: 1) hop to stabilization (10 reps per direction), 2) hop to stabilization and reach (5 reps per direction), 3) unanticipated hop to stabilization (3 reps), 4) progressive single limb stance (3 reps), and 5) progressive single limb stance with eyes closed (3 reps).
  STARS: The STARS intervention will consist of 4 unique sensory-targeted interventions: calf stretching, ankle joint traction, anterior/posterior ankle joint mobilizations, and plantar massage. These four techniques will be applied in the same order for all treatment sessions: 1) 60-second calf stretch, 2) 30-second ankle traction, 3) 30-second mobilization, 4) 2-minute plantar massage, 5) 30-second ankle traction, and 6) 30-second mobilization.
Period: Overall Study
Arm/Group | Balance Training | Balance Training w/ STARS
Started | 12 | 12
Completed | 12 | 12
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Balance Training w/ STARS: Balance Training: This is a 4-week supervised balance training program. During the 4-week program, subjects will complete three 20-25 minute sessions a week for a total of twelve supervised training sessions. Exercises and reps that will be performed per training session will include: 1) hop to stabilization (10 reps per direction), 2) hop to stabilization and reach (5 reps per direction), 3) unanticipated hop to stabilization (3 reps), 4) progressive single limb stance (3 reps), and 5) progressive single limb stance with eyes closed (3 reps).
  STARS: The STARS intervention will consist of 4 unique sensory-targeted interventions: calf stretching, ankle joint traction, anterior/posterior ankle joint mobilizations, and plantar massage. These four techniques will be applied in the same order for all sessions: 1) 60-second calf stretch, 2) 30-second ankle traction, 3) 30-second mobilization, 4) 2-minute plantar massage, 5) 30-second ankle traction, and 6) 30-second mobilization.
- Total: Total of all reporting groups
Arm/Group | Balance Training | Balance Training w/ STARS | Total
Number analyzed (Participants) | 12 | 12 | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 21.3 (1.7) | 21.8 (2.5) | 21.5 (2.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 6 | 14
  Male | 4 | 6 | 10
Region of Enrollment [Number; unit: participants]
  United States | 12 | 12 | 24
Foot and Ankle Ability Measure [Mean (Standard Deviation); unit: % of total questionnaire points] — The Foot and Ankle Ability Measure (FAAM) contains 21 activity related items (max score of 84). Lower percentages (patient's score divided by max score) represent greater disability. The FAAM has been found to be reliable and precise (r=0.89, SEM= 2.1) in people with CAI.
  % of total questionnaire points | 87.1 (8.1) | 86.5 (5.6) | 86.8 (6.9)
Foot and Ankle Ability Measure-Sport [Mean (Standard Deviation); unit: % of total questionnaire points] — The Foot and Ankle Ability Measure- Sports (FAAM-S) contains 8 activity related items (max score of 32). Lower percentages (patient's score divided by max score) represent greater disability. The FAAM-S has been found to be reliable and precise (r=0.87, SEM= 4.5) in people with CAI.
  % of total questionnaire points | 66.2 (12.0) | 72.2 (10.4) | 68.9 (11.4)
Star Excursion Balance Test- Anterior Reach [Mean (Standard Deviation); unit: % of leg length] — To conduct the reach trials, participants placed the test limb in a grid center and kept their hands on their hips. Participants then reached as far as possible in the test direction with the non-test limb. Reach distance was defined as the farthest point that an individual could touch without accepting weight and maintaining balance through the return to a bilateral stance. Reach distance was normalized to the participant's leg length (distance from the anterior superior iliac spine to the ipsilateral medial malleolus). This is a reliable measure of dynamic balance (ICC2,1=0.85-0.96).
  % of leg length | 68.7 (8.3) | 66.2 (6.9) | 67.5 (7.6)
Star Excursion Balance Test- Posteriomedial Reach [Mean (Standard Deviation); unit: % of leg length] — To conduct the reach trials, participants placed the test limb in a grid center and kept their hands on their hips. Participants then reached as far as possible in the test direction with the non-test limb. Reach distance was defined as the farthest point that an individual could touch without accepting weight and maintaining balance through the return to a bilateral stance. Reach distance was normalized to the participant's leg length (distance from the anterior superior iliac spine to the ipsilateral medial malleolus). This is a reliable measure of dynamic balance (ICC2,1=0.85-0.96).
  % of leg length | 79.5 (9.3) | 78.5 (6.7) | 79.0 (8.0)
Star Excursion Balance Test- Posteriolateral Reach [Mean (Standard Deviation); unit: % of leg length] — To conduct the reach trials, participants placed the test limb in a grid center and kept their hands on their hips. Participants then reached as far as possible in the test direction with the non-test limb. Reach distance was defined as the farthest point that an individual could touch without accepting weight and maintaining balance through the return to a bilateral stance. Reach distance was normalized to the participant's leg length (distance from the anterior superior iliac spine to the ipsilateral medial malleolus). This is a reliable measure of dynamic balance (ICC2,1=0.85-0.96).
  % of leg length | 75.7 (12.4) | 72.3 (11.3) | 74.0 (11.7)

OUTCOME MEASURES:

1. Primary Outcome: Balance
Description: Dynamic balance will be assessed with the Star Excursion Balance Test (SEBT). This test requires a person to maintain their balance on a single limb while reaching as far as they can (with their other leg) in 3 different directions (forward, back-left, and back-right).
Time Frame: Balance at 1-day post intervention
Measure: Mean (Standard Deviation); unit: % of leg length
Arm/Group | Balance Training | Balance Training w/ STARS
Number analyzed (Participants) | 12 | 12
% of leg length
  Star Excursion Balance Test: Anterior Reach | 68.7 (8.3) | 66.2 (6.9)
  Star Excursion Balance Test: Posteriomedial Reach | 87.7 (9.0) | 85.5 (8.4)
  Star Excursion Balance Test: Posteriolateral Reach | 83.9 (10.8) | 81.0 (7.44)
Statistical Analysis 1: Comparison: Balance Training vs Balance Training w/ STARS; This analysis examined the change in balance scores from baseline to 1-day post intervention for all three reach distances (Anterior, Posteriomedial, Posteriolateral) using a MANOVA; Test type: Superiority or Other; p = .904, MANOVA

2. Secondary Outcome: Balance
Description: as for outcome 1
Time Frame: Change from baseline balance at 1-week post intervention
Reporting Status: Not Posted

3. Primary Outcome: Self-assessed Disability
Description: 2 questionnaires regarding self-assessed disability during activities of daily living and sport will be completed. The questionnaires will include the Foot and Ankle Ability Measure, and the Foot and Ankle Ability Measure-Sport. The FAAM contains 21 activity related items (max score of 84) while the FAAM-S contains 8 activity related items (max score of 32). Lower percentages (patient's score divided by max score) represent greater disability, and both FAAM and FAAM-S scores have been found to be reliable and precise (r=0.89, SEM= 2.1 and r=0.87, SEM= 4.5, respectively) in people with CAI.
Time Frame: Disability to 1-day post intervention
Measure: Mean (Standard Deviation); unit: % of total questionnaire points
Arm/Group | Balance Training | Balance Training w/ STARS
Number analyzed (Participants) | 12 | 12
% of total questionnaire points
  Foot and Ankle Ability Measure | 89.7 (5.3) | 88.2 (7.9)
  Foot and Ankle Ability Measure- Sport | 76.4 (12.4) | 77.4 (9.6)
Statistical Analysis 1: Comparison: Balance Training vs Balance Training w/ STARS; This analysis examined the change in disability scores from baseline to 1-day post intervention for both disability scores (FAAM, FAAM-S) using a MANOVA; Test type: Superiority or Other; p = .5, MANOVA

4. Secondary Outcome: Self-assessed Disability
Description: 2 questionnaires regarding self-assessed disability during activities of daily living and sport will be completed. The questionnaires will include the Foot and Ankle Ability Measure, and the Foot and Ankle Ability Measure-Sport.
Time Frame: Change from baseline disability at 1-week post intervention
Reporting Status: Not Posted

5. Secondary Outcome: Self-assessed Disability
Description: 3 questionnaires regarding self-assessed disability during activities of daily living and sport will be completed. The questionnaires will include the Ankle Instability Instrument, the Foot and Ankle Ability Measure, and the Foot and Ankle Ability Measure-Sport.
Time Frame: Change from baseline disability at 1-month post intervention
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: During 4 week intervention
Arm/Group | Balance Training | Balance Training w/ STARS
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 0/12 | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No